CLINICAL TRIAL: NCT02597231
Title: Melatonin and Sleep in Preventing Delirium in the Hospital: A Randomized Placebo-controlled Trial
Brief Title: Melatonin and Sleep in Preventing Delirium in the Hospital
Acronym: MELO
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Scripps Health (Other)
Collaborators: Scripps Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: IRB-15-6639
Record Dates: First submitted 2015-10-01; First posted 2015-11-05 (Estimated); Last update posted 2017-10-04 (Actual); Status verified 2017-10

CONDITIONS: Delirium
Keywords: Delirium; Melatonin
MeSH Terms: conditions — Delirium | interventions — Melatonin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Melatonin Group (Experimental): Patients in this group will receive melatonin 3mg orally at 9pm.
  Interventions: Dietary Supplement: Melatonin
- Placebo Group (Placebo Comparator): Patient in this group will receive a matching placebo pill orally at 9pm.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Melatonin — Melatonin is the dietary supplement we are using in delirium prevention.
  Arms: Melatonin Group
Other: Placebo — Patients in this group will receive a matching placebo pill.
  Arms: Placebo Group

SUMMARY:
Recent data suggests that melatonin, a supplement available over the counter, may help prevent delirium in hospitalized patients. The investigators are hypothesizing that melatonin may help in delirium prevention by improving sleep quality and possibly circadian rhythm cycling in patients who are given the supplement. This pilot study involves a randomized placebo-controlled design in which participants will be randomized to receive either melatonin 3mg orally or placebo orally. Participants in both groups will be fitted with wireless actigraphy devices to obtain objective sleep quality, and will also receive a sleep questionnaire each morning to obtain subjective data on their sleep quality overnight. Delirium will be assessed by floor nurses twice daily using the Confusion Assessment Method (CAM).

ELIGIBILITY:
Inclusion Criteria:

* 65-100 years old
* Admitted to Scripps Green Hospital
* Admitted to an Internal Medicine or Medicine Consult Service
* Expected to have a hospital stay of greater than or equal to 48 hours (patients admitted to "inpatient," not "observation," under Medicare guidelines)

Exclusion Criteria:

* Cirrhosis of any etiology
* Admitted for alcohol withdrawal
* Currently taking a 1st or 2nd generation anti-psychotic
* Active delirium (i.e., delirium prior to 1st dose of melatonin)
* Diagnosis of encephalitis
* History of seizure

Ages: 65 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 94 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12-31 (Actual)

PRIMARY OUTCOMES:
Delirium as measured by CAM Assessment | Delirium assessments will be made twice daily (am and pm measurements) throughout the course of the patient's admission, or to the end of a 2 week period of enrollment - whichever comes first.
  Primary outcome is whether patients become delirious, as measured by CAM during their hospital admission.

SECONDARY OUTCOMES:
Objective Sleep Quality, measured by nocturnal sleep duration | nightly, throughout the course of the patient's admission, or to the end of a 2 week period of enrollment - whichever comes first.
  Nocturnal sleep duration will be measured by wireless actigraphy.
Objective sleep quality, measured by number of nighttime wakenings | nightly, throughout the course of the patient's admission, or to the end of a 2 week period of enrollment - whichever comes first.
  We will measure the number of nighttime wakenings using wireless actigraphy.
Objective sleep quality, measured by sleep latency | nightly, throughout the course of the patient's admission, or to the end of a 2 week period of enrollment - whichever comes first.
  We will measure sleep latency (time to fall asleep) using wireless actigraphy.
Subjective sleep quality, measured by Richards-Campbell sleep questionnaire | once daily, throughout the course of the patient's admission, or to the end of a 2 week period of enrollment - whichever comes first.
  Patients will be asked to fill out the Richards-Campbell sleep question, which uses a visual analog scale for 5 questions that are designed to assess a patient's perceived sleep quality.

OTHER OUTCOMES:
Mortality | 6 month
Disposition following hospitalization | 1 day following hospital discharge or at the 2 week time end point of the study.
  We want to determine if the patient is discharged to home, to a post-acute care facility, or to a new type of living facility that was different from their prior living situation.
Subjective sleep quality following hospital discharge. | 6 months following hospital discharge
  Patients will be given an insomnia questionnaire over the phone at 6 months.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas McCarthy, MD, Principal Investigator — Scripps Health
Locations (1):
- Scripps Green Hospital, La Jolla, California, United States

REFERENCES:
- [Derived] Jaiswal SJ, Kang DY, Wineinger NE, Owens RL. Objectively measured sleep fragmentation is associated with incident delirium in older hospitalized patients: Analysis of data collected from an randomized controlled trial. J Sleep Res. 2021 Jun;30(3):e13205. doi: 10.1111/jsr.13205. Epub 2020 Oct 13. PMID 33051948
- [Derived] Jaiswal SJ, McCarthy TJ, Wineinger NE, Kang DY, Song J, Garcia S, van Niekerk CJ, Lu CY, Loeks M, Owens RL. Melatonin and Sleep in Preventing Hospitalized Delirium: A Randomized Clinical Trial. Am J Med. 2018 Sep;131(9):1110-1117.e4. doi: 10.1016/j.amjmed.2018.04.009. Epub 2018 May 3. PMID 29729237